CLINICAL TRIAL: NCT00189020
Title: Effect of 2 Versus 3 Pneumococcal Conjugate Vaccinations Prevnar on Nasopharyngeal Carriage, Transmission and Herd-immunity;a Randomized, Controlled Study
Brief Title: Effect of Two Versus Three Pneumococcal Conjugate Vaccinations
Acronym: MNOES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government); Netherlands Vaccine Institute (Unknown)
Responsible Party: Principal Investigator, Prof Dr EAM Sanders, prof. dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MINOES 01, STEG R05 008; ISRCTN (Registry Identifier: 25571720)
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Streptococcus Pneumoniae Infection
Keywords: pneumococcal conjugate vaccination; nasopharyngeal carriage; herd immunity; antipneumococcal antibodies; respiratory tract infections; National infant vaccination program
MeSH Terms: conditions — Pneumococcal Infections; Respiratory Tract Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2-dose (Experimental): PCV7 at age 2 and 4 months
  Interventions: Biological: PCV7
- 2+1-dose (Experimental): PCV7 at age 2, 4 and 11 months
  Interventions: Biological: PCV7
- Control (No Intervention): Control group

INTERVENTIONS:
Biological: PCV7 — PCV7 at age 2 and 4 months
  Other Names: Prevenar
  Arms: 2-dose
Biological: PCV7 — PCV7 at age 2, 4 and 11 months
  Other Names: Prevenar
  Arms: 2+1-dose

SUMMARY:
Two( 2) or three (3) instead of four vaccinations before the age of 6 months with pneumococcal conjugate vaccine are presumed to protect children against invasive pneumococcal disease like meningitis, at least on the short term till 18-24 months of age. The current hypothesis in this study is 2 or 3 vaccinations will protect against IPD but will not alter pneumococcal nasopharyngeal carriage in infants, and consequently not change pneumococcal transmission and induce no herd-immunity. Furthermore, antibody development and memory may benefit from carriage of vaccine type S. pneumoniae

DETAILED DESCRIPTION:
Two(2 and 4 months) and three vaccinations (2,4 and 11 months) with 7-valent pneumococcal conjugate vaccine Prevnar in infants are presumed to provide about 90% protection against invasive pneumococcal disease (IPD) for vaccine type pneumococci, at least until 18-24 months of age. Licensure of the vaccine however is based on studies with 3 vaccinations before 6 months and a booster vaccination half a year later (3+1 scheme). Cost-effectiveness in national infant vaccination programs (NIPs)is much improved by high herd-immunity effects,as observed in the USA after licensure of Prevnar in 2000, both for IPD and AOM. However, overall pneumococcal carriage reduction (and nasopharyngeal replacement) has not been assessed in studies with reduced doses. With reduced carriage reduction, effects on respiratory tract infections and herd immunity may be significantly less.

The primary aim of the current study is to compare effect of 2-doses (at ages 2 and 4 months) with a 3-doses scheme(2+1, at 2, 4 and 11 months) on nasopharyngeal pneumococcal carriage and replacement and family transmission(sibs and caregivers), in order to allow modelling for herd-immunity.

The secondary aim is to determine the effect of a reduced doses scheme on serum antipneumococcal antibody levels at the age of 12 and 24 months.

A third aim is to determine antipneumococcal antibody levels and memory B-cell development after booster vaccination at 24 months of age, after 2 or 2+1 doses and compare these with a first vaccination at 24 months of age.

Opportunities are the determination of nasopharyngeal colonizing pneumococci in unvaccinated infants in the Netherlands before implementation of Prevnar in the NIP, evaluation of replacing pneumococci in the nasopharynx after vaccinations and analysis of effects on other colonizing bacteria like H.influenzae, M. catarrhalis and S.aureus. Furthermore, the relation between colonizing pneumococci and serotypes causing IPD in the Netherlands can be evaluated.

Methods : 1000 infants and families will be included in a randomized,controlled study with 3 interventions groups

1. Prevnar at 2 and 4 months
2. Prevnar at 2, 4 and 11 months
3. Prevnar at 24 months (controls)

The children will be followed until 2 years of age with nasopharyngeal swabs for bacterial culture before the first vaccination, at 6, 12, 18 and 24 months of age. One sibling and one parent/caregiver will be swabbed when the infant is 12 and 24 months. Blood for antibody determination will be obtained from 80 children of groups 1 and 2, and from 30 children in the control group. Questionnaires on health and respiratory infections and antibiotic prescription for RTI will be obtained.

At 24 months of age, all children of groups 1 and 2 will be offered a booster vaccination. Antibody levels will be measured before and 4 weeks after this vaccination at 2 years of age in a subset of 80 children per group and compared with 80 children who received a first vaccination at 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants eligible for participation in the national infant vaccination program in the Netherlands

Exclusion Criteria:

exclusion from the national vaccination program because of the presence of

* a medical condition requiring treatment that can interfere with the effect of vaccinations
* known or suspected allergy to components of the pneumococcal conjugate vaccine
* known or suspected immunodeficiency disease
* previous treatment with plasma or immunoglobulins
* previous vaccinations other than hepatitis B vaccinations
* coagulation disorders

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1005 (Actual)
Dates: Start 2005-06; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Nasopharyngeal bacterial (pneumococcal) colonization at 6 weeks, 6, 12, 18 and 24 months in infants and at 12 and 24 months of family members | duration of study, 23 months per subject
transmission to family members( sib, caregiver) | at infants age of 12 and 24 months

SECONDARY OUTCOMES:
anti-pneumococcal antibody levels at 12 and 24 months of age | 23 months
antibody levels and B-memory cells after vaccination at 24 months | 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth A. M. Sanders, MD, PhD, Principal Investigator — UMC Utrecht

REFERENCES:
- [Derived] Biesbroek G, Tsivtsivadze E, Sanders EA, Montijn R, Veenhoven RH, Keijser BJ, Bogaert D. Early respiratory microbiota composition determines bacterial succession patterns and respiratory health in children. Am J Respir Crit Care Med. 2014 Dec 1;190(11):1283-92. doi: 10.1164/rccm.201407-1240OC. PMID 25329446
- [Derived] Biesbroek G, Bosch AA, Wang X, Keijser BJ, Veenhoven RH, Sanders EA, Bogaert D. The impact of breastfeeding on nasopharyngeal microbial communities in infants. Am J Respir Crit Care Med. 2014 Aug 1;190(3):298-308. doi: 10.1164/rccm.201401-0073OC. PMID 24921688
- [Derived] Biesbroek G, Wang X, Keijser BJ, Eijkemans RM, Trzcinski K, Rots NY, Veenhoven RH, Sanders EA, Bogaert D. Seven-valent pneumococcal conjugate vaccine and nasopharyngeal microbiota in healthy children. Emerg Infect Dis. 2014 Feb;20(2):201-10. doi: 10.3201/eid2002.131220. PMID 24447437
- [Derived] van Westen E, Rodenburg GD, van Gils EJ, Tcherniaeva I, Berbers GA, Cowell L, Goldblatt D, Rots NY, van den Dobbelsteen GP, Sanders EA. Levels and functionality of antibodies after pneumococcal conjugate vaccine in schedules with different timing of the booster dose. Vaccine. 2013 Dec 2;31(49):5834-42. doi: 10.1016/j.vaccine.2013.09.073. Epub 2013 Oct 10. PMID 24120678
- [Derived] Rodenburg GD, van Gils EJ, Veenhoven RH, Bogaert D, van den Dobbelsteen GP, Berbers GA, Sanders EA. Lower immunoglobulin G antibody responses to pneumococcal conjugate vaccination at the age of 2 years after previous nasopharyngeal carriage of Streptococcus pneumoniae. J Pediatr. 2011 Dec;159(6):965-70.e1. doi: 10.1016/j.jpeds.2011.06.011. Epub 2011 Aug 2. PMID 21813135
- [Derived] van Gils EJ, Hak E, Veenhoven RH, Rodenburg GD, Bogaert D, Bruin JP, van Alphen L, Sanders EA. Effect of seven-valent pneumococcal conjugate vaccine on Staphylococcus aureus colonisation in a randomised controlled trial. PLoS One. 2011;6(6):e20229. doi: 10.1371/journal.pone.0020229. Epub 2011 Jun 10. PMID 21695210
- [Derived] van Gils EJ, Veenhoven RH, Hak E, Rodenburg GD, Keijzers WC, Bogaert D, Trzcinski K, Bruin JP, van Alphen L, van der Ende A, Sanders EA. Pneumococcal conjugate vaccination and nasopharyngeal acquisition of pneumococcal serotype 19A strains. JAMA. 2010 Sep 8;304(10):1099-106. doi: 10.1001/jama.2010.1290. PMID 20823436
- [Derived] van Gils EJ, Veenhoven RH, Hak E, Rodenburg GD, Bogaert D, Ijzerman EP, Bruin JP, van Alphen L, Sanders EA. Effect of reduced-dose schedules with 7-valent pneumococcal conjugate vaccine on nasopharyngeal pneumococcal carriage in children: a randomized controlled trial. JAMA. 2009 Jul 8;302(2):159-67. doi: 10.1001/jama.2009.975. PMID 19584345